CLINICAL TRIAL: NCT02527850
Title: Effect of Low Level Laser Irradiation on Muscle Performance and Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0028-15
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Physical Exertion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment with real laser (Experimental): 10 min irradiation with B-cure soft laser on 3 points of quadriceps muscle.
  Interventions: Device: B-cure laser
- sham laser (Sham Comparator): 10 min irradiation with sham B-cure soft laser on 3 points of quadriceps muscle.
  Interventions: Device: B-cure laser

INTERVENTIONS:
Device: B-cure laser

SUMMARY:
Low level laser therapy (LLLT) was shown to affect muscle performance and fatigue. The aim of this study is to investigated the effect of B-cure laser on muscle performance and recovery after intense exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy physical education students, ages 20-35, light or intermediate skin color

Exclusion Criteria:

musculoskeletal injury to hips or knees in the previous 2 months, use pharmacological agents or nutritional supplements regularly, smokers, physical limitations on completing the exercise tests -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
improvement in muscle power as indicated in 5 repetitions of flexion/extension of the knee using isokinetic dynamometer before and after laser treatment | 1 hour
evaluation of muscle power after induction of muscle fatigue in 5 repetitions of flexion/extension of the knee using isokinetic dynamometer before and after laser treatment | 2 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Wingate Institute, Netanya, Israel